CLINICAL TRIAL: NCT05407467
Title: KurCoSmart Effects on People With Type 2 DM: a Randomized, Open Trial
Brief Title: KurCoSmart Effects on People With Type 2 DM
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitas Sebelas Maret (Other)
Responsible Party: Principal Investigator, Nurhasan Agung Prabowo, M.D., Universitas Sebelas Maret
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: KurCoSmart
Record Dates: First submitted 2022-05-18; First posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Diabetes Mellitus, Type 2; Insulin Resistance; Inflammation; Body Weight
Keywords: curcumin; coconut oil; diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Inflammation; Body Weight; Diabetes Mellitus | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): There is no additional intervention other than subject's standard diabetes treatment
- Interventional Group (Experimental): This group will received additional supplementation of curcumin and virgin coconut oil aside from their standard treatment
  Interventions: Dietary Supplement: Curcumin and virgin coconut oil extract (KurCo Smart)

INTERVENTIONS:
Dietary Supplement: Curcumin and virgin coconut oil extract (KurCo Smart) — we give 2 tablets of curcumin and virgin coconut oil extract thrice a day for 30 days and evaluate the result
  Arms: Interventional Group

SUMMARY:
The investigators aim to evaluate the effect of curcumin and virgin coconut oil extract supplementation on people with type 2 DM, including blood glucose, HbA1c levels, inflammation, body weight and insulin resistance evaluation

DETAILED DESCRIPTION:
The investigators give Kurcosmart supplementation aside from diabetes standard treatment to evaluate its benefits on people with type 2 DM, considering its effect on controlling fasting and prandial blood glucose, reducing HbA1c level, controlling inflammation degree; and repairing insulin resistance

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Type 2 DM
* Signing consent form

Exclusion Criteria:

* Pregnant or breastfeeding
* Multiple organ failure
* History of hypersensitivity reaction to curcumin and virgin coconut oil
* Cancer, renal insufficiency, hematological disease, acute heart failure, chronic liver disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Blood glucose | Change of Blood glucose at 1 months
  Subject's fasting and prandial blood glucose
Inflammation degree | Change of hs-CRP at 1 Months
  Subject's high sensitivity C-reactive protein level
insulin resistance | Change of HOMA IR at 1 Months
  Subject's HOMA IR
HbA1c | Change of HbA1C at 1 Months
  Subject's glycated haemoglobin level

SECONDARY OUTCOMES:
Body Mass Index | Change of BMI at 1 Months
  Subject's height and body weight
Blood Pressure | Change fof blood prssure at 1 Months
  Subject's blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- UNS Hospital, Sukoharjo, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be restricted for this study purpose only